CLINICAL TRIAL: NCT06907732
Title: Fetoscopic Robotic Open Spina Bifida Treatment - a Pilot Feasibility Study
Brief Title: Fetoscopic Robotic Open Spina Bifida Treatment
Acronym: FROST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Tim Van Mieghem, Maternal-Fetal Medicine specialist, Clinician-Investigator, Mount Sinai Hospital, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FROST001
Record Dates: First submitted 2025-02-27; First posted 2025-04-02 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-03

CONDITIONS: Fetal Congenital Abnormalities; Fetoscopy; Fetal Surgery; Robotic Surgical Procedure; Neural Tube Defect; Open Spina Bifida
MeSH Terms: conditions — Neural Tube Defects; Spina Bifida Cystica

STUDY DESIGN:
Intervention Model Description: Exploratory open-label surgical phase 1 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fetoscopic robotic open spina bifida closure (Experimental): Participants in this single study arm will undergo fetoscopic robot-assisted open fetal spina bifida closure.
  Interventions: Procedure: Fetoscopic robotic open spina bifida closure

INTERVENTIONS:
Procedure: Fetoscopic robotic open spina bifida closure — Three 9 mm laparoscopic trocars will be inserted into the uterus after the uterus is exteriorized through a maternal laparotomy. Partial amniotic carbon dioxide insufflation will be done with heated humidified gas. Using a surgical robot, multilayer closure of the lesion will be performed, similar to our current protocol in open fetal spina bifida closure (durapatch, myofascial flap, skin closure).
  Pre- and postoperative management will be similar to our current open fetal surgery protocol. Delivery will be by cesarean section, either when spontaneous labor occurs or at 39 weeks, whichever presents first.

SUMMARY:
Fetal spina bifida is a common birth defect that results in hydrocephalus, motor-, bowel-, bladder- and sexual dysfunction in the child. The condition is progressive in utero. Fetal surgery between 22-26 weeks gestation has been shown to stop the gradual fetal deterioration observed in this disease and improve infant outcomes. Children with spina bifida who have undergone fetal surgery have a lower need for hydrocephalus treatment (80%->40%) and twice the chance to walk independently by the age of 3 years (20%->40%). These benefits are also sustained in the longer term.

The traditional 'open' fetal surgical approach, however, as currently offered clinically at the Ontario Fetal Centre, comes with significant risks: it increases the risk of preterm birth, carries significant maternal morbidity and results in important uterine scarring. The latter comes with a risk of uterine rupture and fetal death both in the index pregnancy and future pregnancies.

To overcome these down sides of open fetal surgery, different centers have attempted a fetoscopic approach to the surgery. Fetoscopy indeed avoids uterine scarring and is likely protective against uterine rupture but is technically complex. This results in long surgical learning curves, poor dissemination of the surgery amongst centers worldwide, longer procedures and suboptimal surgical results which translate in decreased infant benefits - particularly with regards to motor function.

The investigators have developed a fetoscopic robotic approach where they leverage the dexterity of robotic instruments to perform these complex surgeries. The team expects that this will result in easier and faster procedures with better surgical outcomes and therefore fetal benefits comparable to open fetal surgery, while at the same time avoiding the need for hysterotomy.

In this prospective exploratory phase 1 study, the investigators propose to assess the feasibility of such a robotic approach, as developed and trained on a high-fidelity phantom, in 15 patients. The research team will collect maternal and fetal safety and efficacity data to inform later studies.

ELIGIBILITY:
Inclusion Criteria:

* Isolated open fetal spina bifida
* Healthy pregnant patient without risk factors for preterm delivery
* Candidate for open fetal spina bifida surgery.
* Maternal age 18 years or more and able to consent
* Provision of written informed consent to participate in this study
* Gestational age allowing for fetal surgery prior to 26 weeks gestation.

Exclusion Criteria:

* Contraindication for surgery or safe anesthesia due to a severe maternal medical condition, including morbid obesity (BMI >40 kg/m2)
* History of preterm birth, short cervical length, cervical cerclage
* Placenta or vasa previa, invasive placentation
* Inaccessibility of the uterus due to severe maternal obesity, uterine fibroids, bowel or placental superposition
* Major fetal structural or genetic anomalies unrelated to spina bifida, requiring surgery or potentially leading to infant death or severe handicap
* Neural tube defects other than open spina bifida
* Absence of Chiari II malformation on ultrasound or MRI
* Severe fetal kyphosis (>30 degrees)
* Upper lesion level lower than sacral vertebra S1.
* Multiple gestation
* Fetal bleeding disorder (eg. Fetal/neonatal allo-immune thrombocytopenia)
* Maternal infectious disorder which could result in materno-fetal transmission (eg HIV with high viral load)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with successful closure of the fetal spinal defect using a laparotomy-assisted fetoscopic robotic technique | 1 hour postoperatively
  Number of patients who underwent successful closure of the fetal spinal defect in layers using a laparotomy-assisted fetoscopic robotic technique without conversion to hysterotomy.

SECONDARY OUTCOMES:
Number of patients with severe fetal complications | At delivery
  Number of patients with severe fetal complications defined as a composite of intraoperative fetal heart rate decelerations requiring intervention and/or intra- or postoperative fetal death.
Number of patients with severe maternal complications | At delivery
  Number of severe maternal complications defined as a composite outcome including: need for maternal blood transfusion for hemorrhage, placental abruption, chorioamnionitis as assessed on placental pathology, ileus, wound infection or dehiscence, other serious maternal morbidity requiring admission to an intensive care unit, scar dehiscence or rupture at the time of delivery
Number of patients experiencing preterm prelabor rupture of membranes | At delivery
  Incidence of Preterm Prelabor Rupture of Membranes (PPROM). Gestational age at PPROM (in weeks' gestation) will also be recorded.
Number of patients experiencing preterm birth | At delivery
  Gestational age at birth will be recorded in weeks (in weeks) and categorized as <28, <32 and <37 weeks' gestation. Number of patients experiencing preterm birth is number of those delivering prior to 37 weeks' gestation.
Number of patients with a severe neonatal complication | At discharge from Neonatal Intensive Care Unit or 28 days of life whichever comes last
  Number of patient with a severe neonatal complication defined as a composite of either: Neonatal death, death before discharge from the neonatal intensive care unit (NICU) or severe neonatal morbidity defined as the presence of at least one of the following: chronic lung disease, patent ductus arteriosus needing medical therapy or surgical closure, necrotising enterocolitis grade 2 or higher, retinopathy of prematurity stage 3 or higher or severe cerebral injury defined as intraventricular hemorrhage grade 3 or higher or cystic periventricular leukomalacia grade 2 or higher.
Number of infants requiring neonatal spinal scar revision | At 28 days of life
  Number of infants requiring neonatal spinal scar revision within 28 days of birth
Number of infants with reversal of hindbrain herniation | At 28 days of life
  Number of infants with reversal of hindbrain herniation (chiari II malformation) as assessed by MRI during pregnancy or within first 28 days of life.

OTHER OUTCOMES:
Number of patients undergoing cesarean delivery | At delivery
  Mode of delivery will be recorded as cesarean delivery, spontaneous vaginal delivery or assisted vaginal delivery. Number of patients undergoing cesarean delivery will be reported
Infant birthweight | At delivery
  Infant birthweight measured in grams
Number of neonates requiring respiratory support | At discharge from Neonatal Intensive Care Unit
  Number of neonates requiring respiratory support defined as continuous positive airway pressure (CPAP) or invasive ventilation.
Duration of Neonatal Intensive Care Unit Stay | At discharge from Neonatal Intensive Care Unit
  Length of initial neonatal stay in the Neonatal Intensive Care unit, measured in days.

IPD SHARING:
Plan to Share IPD: Yes